CLINICAL TRIAL: NCT01252251
Title: A Phase II Study of RAD001 (Everolimus) and Pasireotide (SOM230) LAR in Patients With Advanced Uveal Melanoma
Brief Title: RAD001 (Everolimus) and Pasireotide (SOM230) LAR in Patients With Advanced Uveal Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-123
Record Dates: First submitted 2010-12-01; First posted 2010-12-02 (Estimated); Results first posted 2017-08-01 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2016-06

CONDITIONS: Uveal Melanoma
Keywords: PASIREOTIDE (SOM230); RAD001 (EVEROLIMUS); eye; 10-123
MeSH Terms: conditions — Uveal Melanoma | interventions — Everolimus; pasireotide; Receptor-Like Protein Tyrosine Phosphatases, Class 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RAD001 and pasireotide LAR (Experimental): This study will be an open-label, single-arm, phase II study of RAD001 and pasireotide LAR.
  Interventions: Drug: RAD001 (Everolimus) and Pasireotide (SOM230) LAR

INTERVENTIONS:
Drug: RAD001 (Everolimus) and Pasireotide (SOM230) LAR — Patients will be treated with SOM-230 (pasireotide) LAR 60mg IM once every 28 days and with RAD001 (Everolimus) 10mg PO daily. Each cycle is 28 days. An optional biopsy may be requested required after weeks of therapy. The biopsy may be performed between days 28 and 42.

SUMMARY:
The purpose of this study is to find out what effects, good and/or bad, the drugs everolimus and pasireotide have on the patient and on melanoma. Pasireotide is also called SOM-230. Pasireotide is an experimental drug and is not approved by the Food and Drug Administration. Everolimus is also called RAD001. Everolimus is approved for use in the U.S. for kidney cancer. Everolimus is not approved for treatment of melanomas, but early studies show that it may help some patients with melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed metastatic uveal melanoma.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as > or = to 20 mm with conventional techniques or as > or = to 10 mm with spiral CT scan.
* Patients may have had any number of prior therapies, but cannot have previously been treated with a somatostatin analogue or an mTOR inhibitor. At least 3 weeks must have elapsed since the last dose of systemic therapy. At least 6 weeks must have elapsed if the last regimen included BCNU or mitomycin C. At least 3 months must have elapsed if the last regimen included an anti-CTLA4 antibody. If the last regimen included an anti-CTLA4 antibody, radiographic disease progression since this therapy must be documented.
* Age > or = to 18 years. Because no dosing or adverse event data are currently available on the use of RAD001 and SOM230 in patients <18 years of age, children are excluded from this study but will be eligible for future pediatric trials, if applicable.
* Life expectancy of greater than 3 months.
* ECOG performance status 0 or 1.
* Patients must have normal organ and marrow function as defined below:
* leukocytes > or = to 3,000/mcL
* absolute neutrophil count > or = to 1,500/mcL
* platelets > or = to 100,000/mcL
* hemoglobin > or = to 9.0 g/dL not requiring transfusions within the past 2 weeks
* total bilirubin < 1.5 X institutional upper limit of normal
* AST(SGOT)/ALT(SGPT) ≤ 2.5 X institutional upper limit of normal
* Creatinine ≤ 1.5 X institutional upper limit of normal or creatinine clearance less than 60 ml/min
* Fasting serum cholesterol ≤300 mg/dL OR ≤7.75 mmol/L AND fasting triglycerides ≤ 2.5 x ULN. NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication.
* INR ≤1.5. (Anticoagulation is allowed if target INR ≤ 1.5 on a stable dose of warfarin or on a stable dose of LMW heparin for >2 weeks at time of study initiation).
* Women of childbearing potential must have a negative serum pregnancy test within 14 days of the administration of the first study treatment. Women must not be lactating. Both men and women of childbearing potential must be advised of the importance of using effective birth control measures during the course of the study. Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study.
* Ability to understand and the willingness to sign a written informed consent document.
* Evidence of disease progression, as determined by the investigator.

Exclusion Criteria:

* Patients may not be receiving any other investigational agents.
* Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases. Treated brain metastases must have been stable for at least 2 months.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to RAD001 or SOM230.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or bleeding, severely impaired lung function, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because RAD001 and SOM230 are agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants, breast-feeding should be discontinued.
* Patients with the presence of active or suspected acute or chronic uncontrolled infection or with a history of immunocompromise, including a positive HIV test result (ELISA and Western blot). The safety of a potentially immunosuppressive drug like everolimus is not proven in patients with HIV. HBV DNA and HCV RNA PCR testing are required at screening for all patients with a positive medical history based on risk factors and/or confirmation of prior HBV/HCV infection (see Section 8.0 and hepatitis B/C risk factor screening form.
* Baseline QTc > 450 ms.
* Patients with risk factors for torsades de pointes, including uncorrected hypokalemia, uncorrected hypomagnesemia, family history of long QT syndrome, clinically significant/symptomatic bradycardia, high-grade AV block, autonomic neuropathy (including that caused by diabetes or Parkinson's disease, uncontrolled hypothyroidism, cirrhosis, or the use of concomitant medications known to prolong the QT interval.
* Patients with a history of syncope, family history of idiopathic sudden death, a history of sustained or clinically significant cardiac arrhythmias, symptomatic congestive heart failure (NYHA Class III or IV), unstable angina pectoris, sustained ventricular tachycardia, ventricular fibrillation, advanced heart block, or a history of acute myocardial infarction within the six months preceding enrollment .
* No concomitant anti-cancer chemotherapy or other systemic drugs. Palliative radiation therapy will be allowed as long as the patient meets all other eligibility criteria.
* Refractory nausea and vomiting, chronic gastrointestinal diseases (e.g. inflammatory bowel disease), or significant bowel resection that would preclude adequate absorption.
* Chronic treatment with systemic steroids or another immunosuppressive agent.
* Patients should not receive immunization with attenuated live vaccines during study period or within 1 week of study entry. Close contact with those who have received attenuated live vaccines should be avoided during treatment with RAD001. Examples of live vaccines include intranasal influenza, measles, mumps, rubella, oral polio, BCG, yellow fever, varicella and TY21a typhoid vaccines.
* Patients with prior or concurrent malignancy except for the following: adequately treated basal cell or squamous cell skin cancer, or other adequately treated in situ cancer, or any other cancer from which the patient has been disease free for five years.
* Patients with a fasting plasma glucose > 1.5 ULN. Note: At the principle investigator's discretion, non-eligible patients can be re-screened after adequate medical therapy has been instituted.
* Patients with symptomatic cholelithiasis.
* Patients who have a history of alcohol or drug abuse in the 6 month period prior to receiving treatment with pasireotide or RAD001.
* History of liver disease, such as cirrhosis or chronic active hepatitis B and C.
* Presence of Hepatitis B surface antigen (HbsAg).
* Presence of Hepatitis C antibody test (anti-HCV).
* History of, or current alcohol misuse/abuse within the past 12 months.
* Known gallbladder or bile duct disease, acute or chronic pancreatitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Postow, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual 11/30/2010, Protocol Closed to Accrual 8/11/2015, Primary Completion Date 6/13/2016, Recruitment location is the medical clinic
Period: Overall Study
Arm/Group | RAD001 and Pasireotide LAR
Started | 14
Completed | 13
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | RAD001 and Pasireotide LAR
Number analyzed (Participants) | 14
Age, Continuous [Median (Full Range); unit: years] | 61 [41 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Response (CR)
Description: For patients with metastatic uveal melanoma treated with RAD001 and pasireotide LAR.
Time Frame: at 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | RAD001 and Pasireotide LAR
Number analyzed (Participants) | 13
Participants
  Participants Evaluated | 13
  Complete Response | 0

2. Primary Outcome: Number of Participants With Partial Response (PR)
Description: For patients with metastatic uveal melanoma treated with RAD001 and pasireotide LAR.
Time Frame: at 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | RAD001 and Pasireotide LAR
Number analyzed (Participants) | 13
Participants
  Participants Evaluated | 13
  Partial Response | 0

3. Primary Outcome: Number of Participants With Stable Disease (SD)
Description: For patients with metastatic uveal melanoma treated with RAD001 and pasireotide LAR.
Time Frame: at 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | RAD001 and Pasireotide LAR
Number analyzed (Participants) | 13
Participants | 7

4. Secondary Outcome: Median Progression Free Survival(PFS)
Time Frame: Up to 3 years
Measure: Median (Full Range); unit: weeks
Arm/Group | RAD001 and Pasireotide LAR
Number analyzed (Participants) | 13
weeks | 16 [7 to 23]

5. Secondary Outcome: Safety and Toxicity in This Patient Population.
Description: Safety assessments will consist of monitoring and recording all adverse events, including serious adverse events, the regular monitoring of hematology (including glycosylated hemoglobin and coagulation parameters), blood chemistry (including fasting glucose, thyroid function tests, GH, IGF-1 and prolactin), urinalysis, regular monitoring of vital signs, echocardiography, ECGs, and body weight. Toxicity will be assessed using the NCI-CTC for Adverse Events, version 4.0 (CTCAEv4.0,
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | RAD001 and Pasireotide LAR
Number analyzed (Participants) | 13
Participants
  At least 1 dose reduction due to toxicity | 7
  No dose reduction due to toxicity | 6

6. Secondary Outcome: Median Overall Survival (OS)
Time Frame: Up to 3 years
Measure: Median (Full Range); unit: months
Arm/Group | RAD001 and Pasireotide LAR
Number analyzed (Participants) | 13
months | 11 [4.5 to 28.5]

ADVERSE EVENTS:
Time Frame: 28 weeks
Arm/Group | RAD001 and Pasireotide LAR
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 6/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RAD001 and Pasireotide LAR (N=13)
Abdominal pain (Gastrointestinal disorders) | 1
Acute kidney injury (Hepatobiliary disorders) | 2
Dizziness (Nervous system disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Lung infection (Infections and infestations) | 1
Mucositis oral (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RAD001 and Pasireotide LAR (N=13)
Hyperglycemia (Metabolism and nutrition disorders) | 13
Cholesterol high (Investigations) | 11
Hypertriglyceridemia (Metabolism and nutrition disorders) | 11
Hyponatremia (Metabolism and nutrition disorders) | 9
White blood cell decreased (Investigations) | 9
CPK increased (Investigations) | 8
Diarrhea (Gastrointestinal disorders) | 8
Platelet count decreased (Investigations) | 8
Mucositis oral (Gastrointestinal disorders) | 7
Hypophosphatemia (Metabolism and nutrition disorders) | 6
Alkaline phosphatase increased (Investigations) | 5
Nausea (Gastrointestinal disorders) | 5
Neutrophil count decreased (Investigations) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Fatigue (General disorders) | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 4
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 3
Hypokalemia (Metabolism and nutrition disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Serum amylase increased (Investigations) | 3
Constipation (Gastrointestinal disorders) | 2
Dizziness (Nervous system disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Headache (Nervous system disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 2
Lipase increased (Investigations) | 2
Non-cardiac chest pain (General disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Anal mucositis (Gastrointestinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Blurred vision (Eye disorders) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Creatinine increased (Investigations) | 1
Dry mouth (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Fever (General disorders) | 1
Hot flashes (Vascular disorders) | 1
Insomnia (Psychiatric disorders) | 1
Lymphocyte count decreased (Investigations) | 1
Oral pain (Gastrointestinal disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes